CLINICAL TRIAL: NCT04949763
Title: Reliability and Validity of the International Standards for Neurological Classification of Spinal Cord Injury in Patients With Non-traumatic Spinal Cord Lesions
Brief Title: Reliability and Validity of the ISNCSCI in Patients With Non-traumatic Spinal Cord Lesions
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giorgio Scivoletto, MD, PhD, I.R.C.C.S. Fondazione Santa Lucia
Other Study IDs: CE/PROG.838 29-05-20
Record Dates: First submitted 2021-06-22; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Spinal Cord Injuries
Keywords: non traumatic spinal cord injury; ISNCSCI; inter-rater reliability; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: rehabilitation — Patients underwent ususal rehabilitation treatment

SUMMARY:
Aim of the study is to assess the psychometric properties of the International Standards for Neurological Classification of Spinal Cord Injury in subjects with non traumatic lesions.

DETAILED DESCRIPTION:
All patients with non-traumatic SCI consecutively admitted to three Italian SCI centers (IRCCS Fondazione Santa Lucia, Montecatone Rehabilitation Hospital and Istituti Clinici Scientifici Maugeri IRCCS of Pavia) between January 1st 2017 and June 30th 2020 have been prospectively enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* having a non-traumatic SCI
* acute / subacute phase
* any level and severity (ASIA Impairment Scale) of injury
* having a cognitive status that allows collaboration in the exam.

Exclusion Criteria:

* presence of dementia or cognitive decline;
* having a pathology of the peripheral nervous system that may affect the evaluation of ISNCSCI;
* having a multiple sclerosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with non traumatic spinal cord lesions
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Interanational Standards for Neurological Classification of Spinal Cord Injury | 1 year
  standards to evaluate neurological status of subject with spinal cord injury

SECONDARY OUTCOMES:
Spinal Cord Independence Maesure | 1 year
  Outcome measure to evaluate the independence in daily life activities for subjects with spinal cord injury

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be available upon reasonable request

REFERENCES:
- [Background] Rupp R, Biering-Sorensen F, Burns SP, Graves DE, Guest J, Jones L, Read MS, Rodriguez GM, Schuld C, Tansey-Md KE, Walden K, Kirshblum S. International Standards for Neurological Classification of Spinal Cord Injury: Revised 2019. Top Spinal Cord Inj Rehabil. 2021 Spring;27(2):1-22. doi: 10.46292/sci2702-1. No abstract available. PMID 34108832

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT04949763/Prot_SAP_000.pdf